CLINICAL TRIAL: NCT05340959
Title: Evaluating Implant Stability Using Three Devices Osstell®, Periotest® and AnyCheck®: A Prospective Observational Clinical Study.
Brief Title: Evaluating Implant Stability Using Three Devices Osstell®, Periotest® and AnyCheck®
Status: Completed | Type: Observational
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Alamin Yassin Dhahi, Postgraduate Student, University of Baghdad
Other Study IDs: 41193
Record Dates: First submitted 2022-03-27; First posted 2022-04-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patient with single or multiple missing tooth or teeth requiring dental implants: Adult patient with single or multiple missing tooth or teeth requiring dental implants, 40 dental implants will be placed in osteotomy sites based on radiographic findings (CBCT), the primary stability will be measured immediately after implant installation and secondary stability will be measured after 12 weeks .
  Both primary and secondary stability will be measured by three devices:
  1. Osstell®: based on Resonance Frequency Analysis (RFA).
  2. Periotest®: based on damping effect.
  3. AnyCheck®: based on tapping-motion.
  Interventions: Device: Devices: Osstell®, Periotest® and AnyCheck®.

INTERVENTIONS:
Device: Devices: Osstell®, Periotest® and AnyCheck®. — 1. Osstell®: is a device that measure implant stability and based on resonance frequency analysis (RFA). Due to stiffness in the interface between the implant surface and the bone smart peg will vibrates accordingly. the more dense bone the higher stability, the higher frequency and higher Implant Stability Quotient (ISQ) value which is from 1-100.
  2. Periotest®: is a device used to assess osseointegration of dental implants, so it measure implant stability . it is based on damping effect of implant. Showing the measurement digitally on a scale from -8 (low mobility) to 50 (high mobility) PTV units.
  3. AnyCheck®: this is an implant stability meter that measures the stiffness of alveolar bone-implant interface through a tapping motion. Showing the measurement on a scale from 30 (low stability) to 85 (high stability).

SUMMARY:
A prospective observational study guided by the guidelines of Strengthening The Reporting Of Observational Study in Epidemiology (STROBE) in 2014, that will be conducted to evaluate implant stability using three devices; Osstell®, Peiotest® and AnyCheck® and comparing the results.

DETAILED DESCRIPTION:
In this study, 40 dental implants will be installed in osteotomy sites for patients with single or multiple missing tooth or teeth based on radiographic findings (CBCT).

The primary stability will be measured immediately after implant installation using three devices :

1. Osstell : based on resonance frequency analysis (RFA).
2. Periotest: based on damping effect.
3. AnyCheck: based on tapping motion. Secondary stability will be measured after 12 weeks using the same devices mentioned above.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients over 18 years of either gender, having single or multiple missing teeth in the maxilla and/or mandible.
2. Patient with adequate vertical bone height and width for implant placement based on preoperative radiographic findings (CBCT).
3. Ability to tolerate conventional surgical and restorative procedures.
4. Patients who are willing to comply with the study and give their consent.

Exclusion Criteria:

1. Active infection or inflammation in the implant zone.
2. Presence of any uncontrolled systemic diseases.
3. Patients with a history of radiotherapy to the head and neck.
4. Any patient requires advanced and complicated surgical techniques such as sinus lift and bone graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults with missing one or more tooth or teeth seeking for dental implant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Implant stability measured by Osstell®. | Changes in implant stability from baseline value measured immediately after implant installation (primary stability) and after 12 weeks (secondary stability).
  Implant stability will be measured by:
  Osstell® (RFA) that is measured by Implant Stability Quotient (ISQ) Value.
Implant stability measured by Periotest®. | Changes in implant stability from baseline value measured immediately after implant installation (primary stability) and after 12 weeks (secondary stability).
  Implant stability will be measured by:
  Periotest® (damping effect) that is measured by Periotest Value (PTV).
Implant stability measured by AnyCheck®. | Changes in implant stability from baseline value measured immediately after implant installation (primary stability) and after 12 weeks (secondary stability).
  Implant stability will be measured by:
  AnyCheck® (tapping-motion) that is measured by Initial Stability Test (IST) Value.
Correlation between values obtained by the devices | Changes in implant stability from baseline value measured immediately after implant installation (primary stability) and after 12 weeks (secondary stability).
  Correlation between values obtained by:
  1. Osstell® (RFA): measured by Implant Stability Quotient (ISQ) Value.
  2. Periotest® (damping effect): measured by Periotest Value (PTV).
  3. AnyCheck® (tapping-motion): measured by Initial Stability Test (IST) Value.

CONTACTS AND LOCATIONS:
Overall Officials: Alamin Y. Dhahi, B.D.S, Principal Investigator — University of Baghdad
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Medical City, Iraq